CLINICAL TRIAL: NCT04685837
Title: Tele-rehabilitation Versus Face-to-face in the Approach to Non-specific Subacute Low Back Pain
Brief Title: New Technologies in the Management of Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexander Achalandabaso (Other)
Responsible Party: Sponsor-Investigator, Alexander Achalandabaso, Physiotherapy doctor, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEID/HU/2020/48
Record Dates: First submitted 2020-12-17; First posted 2020-12-28 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain; Rehabilitation; Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation group (Experimental): The participants randomly assigned to the tele-rehabilitation group will use a computer application to know and execute the exercise protocol. Before starting the protocol, each participant will be assessed by the principal investigator. He will explain how the application works. They will perform 2 sessions of therapeutic exercise for 8 weeks. At the end of the protocol, they will be re-evaluated by the principal investigator.
  Interventions: Other: therapeutic exercise
- Face to face group (Experimental): Participants randomly assigned to the face-to-face group will use the physical therapy clinic to do the exercises controlled by the principal investigator. Before starting the protocol, each participant will be assessed by the principal investigator. He will explain how the protocol works. They will perform 2 sessions of therapeutic exercise for 8 weeks. At the end of the protocol, they will be re-evaluated by the principal investigator.
  Interventions: Other: therapeutic exercise

INTERVENTIONS:
Other: therapeutic exercise — As soon as the study investigators have obtained a significant sample of patients with non-specific sub-acute low back pain, the intervention will begin.
  The principal investigator will perform an individual assessment of the patients. At the end of the assessment, he will randomly distribute them into two groups. Tele-rehabilitation group and face-to-face group.
  On the one hand, the main researcher will explain the application works to the tele-rehabilitation group. For 8 weeks, they have to perform 2 therapy exercise training sessions following the instructions on the application.
  On the other hand, the researcher will explain the protocol to be followed by the group face to face. In addition, he will provide a schedule to follow a correct development of the protocol. Like the tele-rehabilitation group, they will carry out 16 sessions over 8 weeks.
  At the end of the protocol, the principal investigator will perform an individualized assessment of each of the study participants.

SUMMARY:
Lumbopelvic pain represents one of the leading causes of disability and pain in the world population. It is estimated that 84% of the world's population will suffer from lumbar pelvic pain in their lifetime. This high prevalence causes it to be classified as a public health problem.

Traditional primary care measures have failed to reduce the prevalence, recurrences and costs of this pathology. In the search for treatments focused on reducing public spending, the concept of tele-rehabilitation appears. It is a tool, via telematics, that provides knowledge on rehabilitation and education in neurobiology of pain, demonstrated in cardiovascular and respiratory diseases. It has been suggested that the use of this instrument could help improve the patient's quality of life at the biopsychosocial level.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years.
* Non-specific low back pain less than 12 weeks of evolution.
* Knowledge of new information and communication technologies.
* Internet access.

Exclusion Criteria:

* Inflammatory pathologies of the locomotor system.
* Infectious processes.
* Oncological processes.
* Neurodegenerative diseases.
* Pain with neuropathic characteristics.
* Fractures.
* Lack of fluency in Spanish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the SF-12 Questionnaire

SECONDARY OUTCOMES:
Change in Pain perception | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Visual Analog Scale (VAS) from 0 to 10
Change in Disability | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Oswestry Disability Questionnaire
Change in Physical Activity | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Baecke Physical Activity Questionnaire
Change in Kinesiophobia | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Tampa Kinesiophobia Scale (TSK-11) form 11 to 44
Change in Sleep Quality | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Pittsburgh Sleep Quality Index
Change in Catastrophism | Baseline, 2 months (primary timepoint), 3 months after intervention commencement.
  Using the Pain catastrophizing scale from 0 to 56
Change in Lumbar motor control | Baseline, 2 months (primary timepoint).
  Using the Rocking backward test.
Change in Lumbar motor control | Baseline, 2 months (primary timepoint).
  Using the knee extended test.
Change in Intramuscular contraction capacity erector muscles | Baseline, 2 months (primary timepoint).
  Using the Double straight-leg raise test.
Change in Intramuscular contraction capacity erector muscles | Baseline, 2 months (primary timepoint).
  Using the Ito test.
Change in Intramuscular contraction capacity hip flexor muscles | Baseline, 2 months (primary timepoint).
  Using the Hip flexion test supine position and sitting position
Change in Intramuscular contraction capacity extensor flexor muscles | Baseline, 2 months (primary timepoint).
  Using the Hip extension test prone position

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Villatoro, Principal Investigator — University of Jaén
Locations (1):
- Centro de Fisioterapia Villatoro-Luque, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waddell G, Burton AK. Concepts of rehabilitation for the management of low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):655-70. doi: 10.1016/j.berh.2005.03.008. PMID 15949782
- [Background] Macedo LG, Maher CG, Hancock MJ, Kamper SJ, McAuley JH, Stanton TR, Stafford R, Hodges PW. Predicting response to motor control exercises and graded activity for patients with low back pain: preplanned secondary analysis of a randomized controlled trial. Phys Ther. 2014 Nov;94(11):1543-54. doi: 10.2522/ptj.20140014. Epub 2014 Jul 10. PMID 25013000
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Background] Truter P, Russell T, Fary R. The validity of physical therapy assessment of low back pain via telerehabilitation in a clinical setting. Telemed J E Health. 2014 Feb;20(2):161-7. doi: 10.1089/tmj.2013.0088. Epub 2013 Nov 27. PMID 24283249
- [Background] Dario AB, Moreti Cabral A, Almeida L, Ferreira ML, Refshauge K, Simic M, Pappas E, Ferreira PH. Effectiveness of telehealth-based interventions in the management of non-specific low back pain: a systematic review with meta-analysis. Spine J. 2017 Sep;17(9):1342-1351. doi: 10.1016/j.spinee.2017.04.008. Epub 2017 Apr 13. PMID 28412562
- [Background] Palacin-Marin F, Esteban-Moreno B, Olea N, Herrera-Viedma E, Arroyo-Morales M. Agreement between telerehabilitation and face-to-face clinical outcome assessments for low back pain in primary care. Spine (Phila Pa 1976). 2013 May 15;38(11):947-52. doi: 10.1097/BRS.0b013e318281a36c. PMID 23238489
- [Background] Mbada CE, Olaoye MI, Dada OO, Ayanniyi O, Johnson OE, Odole AC, Ishaya GP, Omole OJ, Makinde MO. Comparative Efficacy of Clinic-Based and Telerehabilitation Application of Mckenzie Therapy in Chronic Low-Back Pain. Int J Telerehabil. 2019 Jun 12;11(1):41-58. doi: 10.5195/ijt.2019.6260. eCollection 2019 Spring. PMID 31341546
- [Background] del Pozo-Cruz B, Gusi N, del Pozo-Cruz J, Adsuar JC, Hernandez-Mocholi M, Parraca JA. Clinical effects of a nine-month web-based intervention in subacute non-specific low back pain patients: a randomized controlled trial. Clin Rehabil. 2013 Jan;27(1):28-39. doi: 10.1177/0269215512444632. Epub 2012 May 31. PMID 22653374
- [Background] Peterson S, Kuntz C, Roush J. Use of a modified treatment-based classification system for subgrouping patients with low back pain: Agreement between telerehabilitation and face-to-face assessments. Physiother Theory Pract. 2019 Nov;35(11):1078-1086. doi: 10.1080/09593985.2018.1470210. Epub 2018 May 3. PMID 29723124
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] Cuesta Vargas AI, Rodríguez Moya A. Frecuencia de uso de escalas de dolor, incapacidad fisica y calidad de vida en el estudio de lumbalgia con intervenciones fisioterápicas. Fisioterapia 2008; 30(4), 204-208.
- [Background] Flórez García MT, García Pérez MA, García Pérez F, et al. Adaptación transcultural a la población española de la escala de incapacidad por dolor lumbar de Oswestry. Rehab (Madr). 1995; 29:138-45.
- [Background] Gomez-Perez L, Lopez-Martinez AE, Ruiz-Parraga GT. Psychometric Properties of the Spanish Version of the Tampa Scale for Kinesiophobia (TSK). J Pain. 2011 Apr;12(4):425-35. doi: 10.1016/j.jpain.2010.08.004. PMID 20926355
- [Background] Hita-Contreras F, Martinez-Lopez E, Latorre-Roman PA, Garrido F, Santos MA, Martinez-Amat A. Reliability and validity of the Spanish version of the Pittsburgh Sleep Quality Index (PSQI) in patients with fibromyalgia. Rheumatol Int. 2014 Jul;34(7):929-36. doi: 10.1007/s00296-014-2960-z. Epub 2014 Feb 8. PMID 24509897